CLINICAL TRIAL: NCT01514903
Title: Pharmacokinetics of Sildenafil Following Administration of an Chewable Tablet of Sildenafil Relative to Viagra® Conventional Oral Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-SIL-102
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Erectile Dysfunction
Keywords: anti erectile dysfunction agent
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- viagra,anti-erectile dysfunction agent (Active Comparator)
  Interventions: Drug: viagra
- HIP0908 (Experimental)
  Interventions: Drug: HIP0908

INTERVENTIONS:
Drug: HIP0908 — SINGLE DOSE , CROSS OVER
  Arms: HIP0908
Drug: viagra — single dose, cross over
  Arms: viagra,anti-erectile dysfunction agent

SUMMARY:
This is a single dose open-label comparative pharmacokinetic study to assess the pharmacokinetic characteristics of sildenafil between HIP0908 (chewable tablet) and Viagra (tablet) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 45
* weight : over 55kg and 18.5 < BMI, 25.0
* have to give their consent to participating clinical trial by oneself

Exclusion Criteria:

* has a medical history of hypersensitivity to drug including PDE5 inhibitor and QTc > 430ms or uncontrolled arrhythmia

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUC and Cmax of sildenafil | Pre-dose (0h), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hr post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Sinchon Severance Hospital, Seoul, South Korea